CLINICAL TRIAL: NCT04955444
Title: Optimization of Opioid Discharge Prescriptions Following Thyroid and Parathyroid Surgeries
Brief Title: Opioid Use After Thyroid and Parathyroid Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: University of Houston (Other)
Responsible Party: Principal Investigator, Elsie Rizk, Pharmacy Administrative Specialist in Clinical Research Program Director, Clinical Pharmacy Fellowship in Outcomes Research, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro000023276
Record Dates: First submitted 2021-06-18; First posted 2021-07-08 (Actual); Results first posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2022-10

CONDITIONS: Thyroidectomy; Parathyroidectomy; Opioid Use; Pain, Postoperative
Keywords: Thyroidectomy; Parathyroidectomy; Opioid; Postoperative pain; Multimodal anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The study consists of 2 groups: (1) the historical control group and (2) the post-implementation group. The historical control group includes 160 patients who underwent a thyroidectomy or a parathyroidectomy procedure from January 2018 to December 2019 (20 patients randomly sampled from each quarter prior to bundle implementation). The quality improvement bundle will be implemented at Houston Methodist Hospital in June 2021. The post-implementation group will include the first 80 eligible patients accrued over 4 to 6 months following bundle implementation. An estimated sample size of 80 patients in the post-implementation group and 160 patients in the historical control group will provide 80% power to detect an absolute decrease of 20% in the primary endpoint using a two-sided alpha of 0.05.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Historical control group (No Intervention): The historical control group underwent a thyroidectomy or parathyroidectomy procedure prior to implementation of the quality improvement bundle.
- Post-implementation group (Experimental): The post-implementation group will have a thyroidectomy or parathyroidectomy procedure after bundle implementation and will receive care that is enhanced by the quality improvement bundle.
  Interventions: Other: Quality improvement bundle

INTERVENTIONS:
Other: Quality improvement bundle — The quality improvement bundle consists of (1) patient education, (2) provider education, and (3) EHR enhancements including order sets and best practice alerts.
  Arms: Post-implementation group

SUMMARY:
Unnecessary opioid prescriptions for postoperative pain can increase the risk for new, persistent opioid use and dependence. Published literature suggests that most patients undergoing thyroid or parathyroid surgery can have their pain effectively managed without opioids following hospital discharge. The purpose of this quasi-experimental, quality improvement study is to develop, implement, and measure the impact of a quality improvement bundle that consists of (1) patient education, (2) provider education, and (3) electronic health record (EHR) enhancements. The proportion of patients who receive new opioid discharge prescriptions for pain management following thyroid or parathyroid surgery at Houston Methodist Hospital for up to 6 months following bundle implementation will be compared to a historical control group.

DETAILED DESCRIPTION:
BACKGROUND: New and persistent opioid use after minor and major surgery is common, and the duration of opioid use following surgery is associated with opioid dependence, abuse, and overdose. Most patients undergoing thyroid or parathyroid surgery do not require opioid discharge prescriptions for effective pain management. If opioids are prescribed for these surgeries, up to 7% of patients will use opioids 3 to 6 months after surgery. Previously published quality programs that optimized perioperative multimodal analgesia (MMA) regimens, provider education, patient education, and shared decision making successfully reduced the proportion of patients discharged with opioid prescriptions to less than 5% following thyroid and parathyroid surgery.

STUDY DESIGN: This quasi-experimental, quality improvement study compares opioid discharge prescribing practices before and after implementation of the quality improvement bundle. The quality improvement bundle includes patient education, provider education, and EHR enhancements. Patients who undergo a thyroidectomy or parathyroidectomy procedure will be included in the study. The historical control group includes patients treated prior to bundle implementation. The post-implementation group includes patients treated within 4 to 6 months following bundle implementation. The primary outcome is the proportion of patients who receive new opioid discharge prescriptions at discharge following a thyroidectomy or parathyroidectomy procedure. This outcome excludes the continuation of previous, chronic opioid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing a primary thyroidectomy or parathyroidectomy procedure at Houston Methodist Hospital during the study period. Only index surgeries during the study time frame were included.

Exclusion Criteria:

* Patients with a hospital length of stay after surgery >2 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elsie Rizk, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Brat GA, Agniel D, Beam A, Yorkgitis B, Bicket M, Homer M, Fox KP, Knecht DB, McMahill-Walraven CN, Palmer N, Kohane I. Postsurgical prescriptions for opioid naive patients and association with overdose and misuse: retrospective cohort study. BMJ. 2018 Jan 17;360:j5790. doi: 10.1136/bmj.j5790. PMID 29343479
- [Background] Jena AB, Goldman D, Karaca-Mandic P. Hospital Prescribing of Opioids to Medicare Beneficiaries. JAMA Intern Med. 2016 Jul 1;176(7):990-7. doi: 10.1001/jamainternmed.2016.2737. PMID 27294595
- [Background] Lou I, Chennell TB, Schaefer SC, Chen H, Sippel RS, Balentine C, Schneider DF, Moalem J. Optimizing Outpatient Pain Management After Thyroid and Parathyroid Surgery: A Two-Institution Experience. Ann Surg Oncol. 2017 Jul;24(7):1951-1957. doi: 10.1245/s10434-017-5781-y. Epub 2017 Feb 3. PMID 28160140
- [Background] Ruffolo LI, Jackson KM, Juviler P, Kaur R, Chennell T, Glover DM, Linehan DC, Moalem J. Narcotic Free Cervical Endocrine Surgery: A Shift in Paradigm. Ann Surg. 2021 Aug 1;274(2):e143-e149. doi: 10.1097/SLA.0000000000003443. PMID 31356280
- [Background] Oltman J, Militsakh O, D'Agostino M, Kauffman B, Lindau R, Coughlin A, Lydiatt W, Lydiatt D, Smith R, Panwar A. Multimodal Analgesia in Outpatient Head and Neck Surgery: A Feasibility and Safety Study. JAMA Otolaryngol Head Neck Surg. 2017 Dec 1;143(12):1207-1212. doi: 10.1001/jamaoto.2017.1773. PMID 29049548
- [Background] Militsakh O, Lydiatt W, Lydiatt D, Interval E, Lindau R, Coughlin A, Panwar A. Development of Multimodal Analgesia Pathways in Outpatient Thyroid and Parathyroid Surgery and Association With Postoperative Opioid Prescription Patterns. JAMA Otolaryngol Head Neck Surg. 2018 Nov 1;144(11):1023-1029. doi: 10.1001/jamaoto.2018.0987. PMID 30027221
- [Background] Shindo M, Lim J, Leon E, Moneta L, Li R, Quintanilla-Dieck L. Opioid Prescribing Practice and Needs in Thyroid and Parathyroid Surgery. JAMA Otolaryngol Head Neck Surg. 2018 Dec 1;144(12):1098-1103. doi: 10.1001/jamaoto.2018.2427. PMID 30422170
- [Background] Sada A, Ubl DS, Thiels CA, Cronin PA, Dy BM, Lyden ML, Thompson GB, McKenzie TJ, Habermann EB. Optimizing Opioid-Prescribing Practices After Parathyroidectomy. J Surg Res. 2020 Jan;245:107-114. doi: 10.1016/j.jss.2019.07.039. Epub 2019 Aug 12. PMID 31415931
- [Background] Overton HN, Hanna MN, Bruhn WE, Hutfless S, Bicket MC, Makary MA; Opioids After Surgery Workgroup. Opioid-Prescribing Guidelines for Common Surgical Procedures: An Expert Panel Consensus. J Am Coll Surg. 2018 Oct;227(4):411-418. doi: 10.1016/j.jamcollsurg.2018.07.659. Epub 2018 Aug 14. PMID 30118896
- [Background] Rizk E, Swan JT, Cheon O, Colavecchia AC, Bui LN, Kash BA, Chokshi SP, Chen H, Johnson ML, Liebl MG, Fink E. Quality indicators to measure the effect of opioid stewardship interventions in hospital and emergency department settings. Am J Health Syst Pharm. 2019 Feb 1;76(4):225-235. doi: 10.1093/ajhp/zxy042. PMID 30715186
- [Result] Rizk E, Yuan F, Zheng F, Fink E, Kaur N, Tran AT, Iso T, Mohyuddin NG, Thekdi AA, Jackson GL, Wanat MA, Thornton JD, Swan JT. Optimization of Opioid Discharge Prescriptions Following Thyroid and Parathyroid Surgery. Otolaryngol Head Neck Surg. 2023 Jul;169(1):176-184. doi: 10.1177/01945998221121626. Epub 2023 Jan 29. PMID 36040827

RESULTS

PARTICIPANT FLOW:
Groups:
- Post-implementation Group: The post-implementation group underwent a thyroidectomy or parathyroidectomy procedure after bundle implementation and received care that is enhanced by the quality improvement bundle.
  Quality improvement bundle: The quality improvement bundle consists of (1) patient education, (2) provider education, and (3) EHR enhancements including order sets and best practice alerts.
Period: Overall Study
Arm/Group | Historical Control Group | Post-implementation Group
Started | 160 | 80
Completed | 160 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Historical Control Group | Post-implementation Group | Total
Number analyzed (Participants) | 160 | 80 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (14) | 57 (14) | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 65 | 197
  Male | 28 | 15 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 14 | 35
  Not Hispanic or Latino | 139 | 66 | 205
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 109 | 49 | 158
  Race: Black or African American | 33 | 23 | 56
  Race: Asian | 10 | 6 | 16
  Race: Other | 8 | 2 | 10
Opioid use within 1 week prior to surgery [Count of Participants; unit: Participants] | 8 | 2 | 10
Surgery performed [Count of Participants; unit: Participants]
  Parathyroidectomy | 82 | 39 | 121
  Thyroidectomy | 90 | 46 | 136

OUTCOME MEASURES:

1. Primary Outcome: New Opioid Discharge Prescriptions
Description: Proportion of patients who receive new opioid discharge prescriptions at discharge following a thyroidectomy or parathyroidectomy procedure. This outcome excludes continuation of previous, chronic opioid therapy.
Time Frame: Up to 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Group | Post-implementation Group
Number analyzed (Participants) | 160 | 80
Participants | 128 | 28

2. Secondary Outcome: Opioid Discharge Prescriptions Exceeding 112.5 Oral Morphine Milligram Equivalents (MMEs)
Description: Proportion of thyroidectomy and parathyroidectomy postoperative patients with opioid discharge prescriptions exceeding the recommended dose of 112.5 oral MMEs
Time Frame: Up to 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Group | Post-implementation Group
Number analyzed (Participants) | 160 | 80
Participants | 52 | 8

3. Secondary Outcome: Opioid Discharge Prescriptions Exceeding 5 Days
Description: Proportion of thyroidectomy and parathyroidectomy postoperative patients with opioid discharge prescriptions exceeding 5 days of therapy
Time Frame: Up to 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Group | Post-implementation Group
Number analyzed (Participants) | 160 | 80
Participants | 27 | 5

4. Secondary Outcome: New Opioid Prescriptions From the Surgeon's Office Within 7 Days of Surgery
Description: Proportion of thyroidectomy and parathyroidectomy postoperative patients who receive new opioid prescriptions from the surgeon's office within 7 days of surgery including discharge prescriptions. This outcome excludes continuation of previous, chronic opioid therapy.
Time Frame: Up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Group | Post-implementation Group
Number analyzed (Participants) | 160 | 80
Participants | 0 | 0

5. Secondary Outcome: Opioid Prescriptions Exceeding 50 Oral MMEs/Day When New Discharge Prescriptions Are Added to Existing Opioid Therapy
Description: Proportion of thyroidectomy and parathyroidectomy postoperative patients with opioid prescriptions exceeding 50 oral MMEs/day when new, postoperative discharge prescriptions are added to existing opioid therapy
Time Frame: Up to 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Group | Post-implementation Group
Number analyzed (Participants) | 160 | 80
Participants | 9 | 0

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study
Arm/Group | Historical Control Group | Post-implementation Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT04955444/Prot_SAP_000.pdf